CLINICAL TRIAL: NCT07296029
Title: Cerebral Oxygenation and Neurological Outcomes FOllowing CriticAL Illness-2 (CONFOCAL-2) Interventional Pilot Study
Brief Title: CONFOCAL-2 Interventional Pilot Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Gordon Boyd, Clinician-Scientist, Queen's University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 6033269
Record Dates: First submitted 2025-03-26; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Critical Illness; Respiratory Failure; Shock; Delirium
Keywords: cerebral oximetry; near-infared spectroscopy; neurocognitive; post-ICU syndrome; precision medicine
MeSH Terms: conditions — Critical Illness; Respiratory Insufficiency; Shock; Delirium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autoregulation-based precision blood pressure management (Experimental): Blood pressure maintenance based on cerebral oximetry autoregulation measurement.
  Interventions: Drug: Autoregulation-based precision blood pressure management

INTERVENTIONS:
Drug: Autoregulation-based precision blood pressure management — Blood pressure maintenance based on cerebral oximetry autoregulation measurement. Blood pressure is raised or lowered via norepinephrine (dose range 1-10 mcg/min) and labetalol (dose range 0-2 mg/min), respectively, to match the researched blood pressure targets.

SUMMARY:
This study is designed to assess the feasibility of identifying and administering individualized blood pressure targets early critical illness. Recent literature suggests that individualized targets adapted to cerebral perfusion and autoregulation capacity may improve patient outcomes. In this study, cerebral autoregulation capacity is assessed by simultaneous trending of near-infared spectroscopy and arterial blood pressure for 24 hours, within patients' first 2 days in the ICU. The investigators will assess the feasibility of identifying patients' personal targets, then treating patients according to their personal targets for 48 hours. Clinical outcomes explored will include delirium.

ELIGIBILITY:
Inclusion Criteria:

1. Admitted to a critical care unit requiring one or more of the following:

   1. Respiratory failure requiring invasive mechanical ventilation with an expected duration >24 hours or
   2. Shock of any etiology. Shock is defined by the need for one of the following vasopressors/inotropes: i. Dopamine ≥7.5 mcg/kg/min, ii. Dobutamine ≥5 mcg/kg/min, iii. Norepinephrine ≥5 mcg/min, iv. Phenylephrine ≥75 mcg/min, v. Epinephrine at any dose, vi. Milrinone at any dose (if used in conjunction with another agent), vii. Vasopressin ≥0.03 u/min (if used in conjunction with another agent)
2. Presence of an arterial line

Exclusion Criteria:

1. Admission to the ICU > 24 hours
2. Life expectancy <24 hours
3. Primary central nervous system admitting diagnosis (e.g. traumatic brain injury, stroke, subarachnoid haemorrhage, cardiac arrest).
4. Pregnancy
5. Any reason that the subject may not be able to participate in the follow up assessments (i.e. limb amputation, paresis, neuromuscular disorders)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2022-07-29 (Actual); Primary Completion 2025-02-08 (Actual); Study Completion 2025-02-08 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | From period of study start to finish, an average of one year.
  Target recruitment rate = 1 patient/month
Determine optimal mean arterial pressure target (MAPopt) | For 24 hours after enrollment
  Aim to determine MAPopt in >75% of patients within the first 24 hours
Maintain MAP within MAPopt range | for 24-72 hours after enrolment
  Aim to maintain patients in MAPopt range for >90% of the time for 48 hours

SECONDARY OUTCOMES:
Correlation between delirium and cerebral autoregulation | Up to day 30 after ICU admission or the day of patient discharge
  Patients will be assessed daily for delirium throughout their entire hospital stay (ICU and ward; up to day 30) using a validated screening tool; the Confusion Assessment Method (CAM)-ICU while in ICU, and the Confusion Assessment Method (CAM) while on the ward. Trained researchers will administer the CAM-ICU once daily, at a time that is convenient for the patient, their family, and the medical team directing their care. The ICU discharge day will be considered to be the day that the attending writes orders to discharge to avoid the influence of delayed ICU discharge because of the lack of ward beds. We will calculate the correlation between the proportion of time spent with dysfunctional cerebral autoregulation and the duration of time with delirium.
Correlation between delirium and time outside MAPopt | Up to day 30 after ICU admission or the day of patient discharge
  Patients will be assessed daily for delirium throughout their entire hospital stay (ICU and ward; up to day 30) using a validated screening tool; the Confusion Assessment Method (CAM)-ICU while in ICU, and the Confusion Assessment Method (CAM) while on the ward. Trained researchers will administer the CAM-ICU once daily, at a time that is convenient for the patient, their family, and the medical team directing their care. The ICU discharge day will be considered to be the day that the attending writes orders to discharge to avoid the influence of delayed ICU discharge because of the lack of ward beds. We will calculate the correlation between the proportion of time spent with dysfunctional cerebral autoregulation and the duration of time with delirium.
Exploratory short-term delirium outcomes | Up to day 30 after ICU admission or the day of patient discharge
  Patients will be assessed daily for delirium throughout their entire hospital stay (ICU and ward; up to day 30) using a validated screening tool; the Confusion Assessment Method (CAM)-ICU while in ICU, and the Confusion Assessment Method (CAM) while on the ward. Trained researchers will administer the CAM-ICU once daily, at a time that is convenient for the patient, their family, and the medical team directing their care. The ICU discharge day will be considered to be the day that the attending writes orders to discharge to avoid the influence of delayed ICU discharge because of the lack of ward beds. We will calculate the correlation between the proportion of time spent with outside of MAPopt and the duration of time with delirium.

CONTACTS AND LOCATIONS:
Locations (1):
- Kingston Health Sciences Center, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
We are open to sharing individual participant data that underlie the results reported in this article after deidentification (text, tables, figures, appendices). Data sharing would be available to interested researchers for IPD meta-analysis or other research aims for which IPD is necessary. Proposals should be directed to study contact Dr. Gordon Boyd at Gordon.Boyd@kingstonhsc.ca. To gain access, data requestors will need to sign a data access agreement.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication
Access Criteria: Researchers who provide a methodologically sound proposal and received ethics approval for their proposal